CLINICAL TRIAL: NCT03324035
Title: Treatment of Neuropathic Pain in Leprosy: a Randomized Double Blind Controlled Study
Brief Title: Treatment of Neuropathic Pain in Leprosy
Acronym: AmyNeLe
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Cristália Produtos Químicos Farmacêuticos Ltda. (Industry)
Responsible Party: Principal Investigator, Daniel Ciampi Araujo de Andrade, MD, PhD, Principal Investigator, Pain Center coordinator, Department of Neurology, University of Sao Paulo, São Paulo, Brazil, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AmyNeLe
Record Dates: First submitted 2017-06-14; First posted 2017-10-27 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Pain, Neuropathic; Leprosy; Leprosy Neuropathy; Amitriptyline
MeSH Terms: conditions — Neuralgia; Leprosy | interventions — Amitriptyline; Tramadol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental): Patients on this arm will receive amitriptyline on flexible doses, starting from 25mg (1 capsule) and titrated to 50mg (2 capsules) or 75mg (3 capsules), based on brief pain inventory (BPI) questionnaire, applied weekly for 3 consecutive weeks. All patients will receive tramadol as a supportive drug for the treatment of neuropathic pain, they are instructed to take 50mg every 8 hours, if pain present.
  Interventions: Drug: Amitriptyline; Drug: Tramadol
- Placebo (Placebo Comparator): Patients on this arm will receive placebo on flexible doses, starting from 1 capsule and titrated to 2 capsules or 3 capsules, based on brief pain inventory (BPI) questionnaire, applied weekly for 3 consecutive weeks. All patients will receive tramadol as a supportive drug for the treatment of neuropathic pain, they are instructed to take 50mg every 8 hours, if pain present.
  Interventions: Drug: Placebo oral capsule; Drug: Tramadol

INTERVENTIONS:
Drug: Amitriptyline — Administer amitriptyline on flexible doses variating from 25mg to 75mg, with backup of tramadol, and evaluate the reduction of the pain based on the Brief Pain Inventory Questionnaire.
  Arms: Treatment
Drug: Placebo oral capsule — Administer amitriptyline on flexible doses variating from 1 to 3 capsules, with backup of tramadol, and evaluate the reduction of the pain based on the Brief Pain Inventory Questionnaire.
  Arms: Placebo
Drug: Tramadol — Administer to both arms on "as needed" scheme, to a maximum of 150mg/day.

SUMMARY:
Despite large efforts to eradicate leprosy, this curable mycobacterial infection still affects 250,000 new individuals annually. Half of the globe's leprosy patients live in Brazil and India. In 2013, 33,033 new leprosy cases diagnosed in Brazil, with an average incidence of 1.05 cases / 10 000 inhabitants. Recently a new concept of care after cure has called attention for severe pain in previously treated patients, particularly, neuropathic pain. Even so, until now no single drug has been studied for the treatment of pain in this patients, and the use of drugs is based on the study of other diseases. We designed the first placebo-controlled, double blinded randomized trial in the use of flexible-dose amitriptyline (tricyclic antidepressant) for the treatment of neuropathic pain related to leprosy

DETAILED DESCRIPTION:
Despite large efforts to eradicate leprosy, this curable mycobacterial infection still affects 250,000 new individuals annually. Half of the globe's leprosy patients live in Brazil and India. In 2013, 33,033 new leprosy cases diagnosed in Brazil, with an average incidence of 1.05 cases / 10 000 inhabitants. Most new cases occur in economically restricted regions of the world, but because at least 5% of the general population is genetically susceptible to the causative agent, new cases may occur anywhere worldwide. This is especially true in times of high human geographic dislocation. Thus, leprosy should rank among the differential diagnosis list of general practitioners and specialists treating skin and peripheral nerve disorders even in non-endemic areas.

Mycobacterium leprae is an obligatory intracellular bacterium that invades macrophages and Schwann cells. Although myelinating Schwann cells are relatively resistant to invasion, viable M. leprae cause marked myelin destruction and lead to secondary neuronal phenotypic changes, degeneration, and nerve dysfunction.

Leprosy patients have historically been characterized by cutaneous insensibility in body areas of deformity, and the presence of pain in these patients has been neglected for a long time. It has only been recently acknowledged that leprosy can be associated with pain in general and neuropathic pain in particular. Leprosy patients frequently experience neuropathy in wide areas of the body, which may or may not present with pain. When pain exists, it may be acute or chronic, neuropathic or inflammatory. Leprosy has different clinical presentations (according to the host's innate immune response) that range from localized skin lesions and adjacent intra-epidermal nerve fiber injury to widespread neuropathy distributed in large areas of low body-surface temperature. Neuropathic pain in leprosy may affect 11-22% of patients, and up to 56% of those with chronic pain. Importantly, more than 85% of patients with leprosy-related neuropathic pain developed it after the end of the antimicrobial treatment period. This means that the majority of patients who developed neuropathic pain did so after they were formally cured of the disease, and, in many cases, discharged from medical assistance. Therefore, pain in leprosy can also be inserted as part of the "care after cure" program initiative, along with stigma, deformity and incapacity management strategies.

In recent years several easy-to use screening tools have been developed to screen for neuropathic pain in leprosy patients, such as the douleur neuropathique-4 (DN-4) and others. These tools allow for the rapid (usually 20 seconds to administer) and reliable (high sensitivity) assessment of pain in leprosy patients.

Additionally, very few reports have described he effects of treatment used for neuropathic pain in these patients, and no clinical trials have been conducted for this specific condition to date. One could argue that leprosy patients with neuropathic pain should respond to usual drugs such as tricyclic antidepressants and anticonvulsants (and they usually do), but the selection of the appropriate treatment regimen, the proper timing of treatment initiation and the most cost-effective drug is not an obvious task. Also, and very important, the lack of formal evidence-based data attesting the efficacy of tricyclics and anticonvulsants for the treatment of leprosy associated neuropathic pain hampers further a wider availability of these drugs in economically-restricted areas. All these limitations can be overcome if the current scientific interest in pain in leprosy is maintained and the present high-level research in the area continues to grow similarly to the previous decades.

Here we designed the first placebo-controlled, double blinded randomized trial in the use of flexible-dose amitriptyline (tricyclic antidepressant) for the treatment of neuropathic pain related to leprosy. This study is currently approved by our local Ethics Review Board (CAAE: 45393415.9.0000.0068) and has stared the recruitment phase on March 2017.

Recruitment time will be extended by 12 months due to dropouts related to the Covid pandemic. We have had dropouts due to a few patients developing covid and also due to patients having fear to become infected while attending hospital visits."

ELIGIBILITY:
Inclusion Criteria:

* Presence of spontaneous pain of medium intensity in the last 24 hours with a minimum value of 4 in 10 on a numerical scale, with a maximum of 10 points (summed pain questionnaire)
* Duration of pain of at least 6 months
* Presence of neuropathic pain "pure" or of clearly dominant character (no other pain, or pain associated unimportant)
* Pain due to leprosy confirmed by clinical examination and / or appropriate electrophysiological examination
* Ability to properly understand the Portuguese language, being able to understand the methodology of the study and questionnaires
* Having provided their consent in writing of their participation in the study

Exclusion Criteria:

* Linked to the disease in study:
* Neuropathic pain from other causes that not Hansen's disease (Diabetes, HIV, and after chemotherapy);
* Linked to the treatment:
* Hypersensitivity to amitriptyline and tramadol;
* Ongoing treatment with monoamine oxidase inhibitors (MAOIs);
* Cardiac and ophthalmologic disorders that contraindicate the use of amitryptiline;
* Pregnant or nursing women, or even women of childbearing age without the use of contraceptives.
* General
* Other pain with intensity higher then the neuropathic one;
* Ant other condition that may interfere with the evaluation of the study;
* Patients who have not given or signed the informed consent form;
* Incorrectly completion of the self-assessment of pain notebook in the period between inclusion and randomization (at least 4 scores in 7 days);
* Patients who can't be followed on a regular basis or that miss the appointments (we will give a 7 day tolerance for each appointment);
* Documented abuse of psychoactive drugs or alcohol;
* History of past or actual psychosis;
* Actual diagnosis of major depression following the DSM-IV criteria;
* Language and cognitive deficits that are capable of interfering with the understanding of the study;
* Patients not affiliated with a social security scheme (beneficiary or recipient);
* Patients who refuses to sign or are unable to understand the informed consent, under guardianship;
* Participation in other research protocol involving the use of any medication during the 30 days preceding the inclusion in the project.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain intensity of 30% from baseline measured by verbal analog scale (VAS) | 63 days (9 weeks)
  To evaluate the analgesic effect of amitriptyline in flexible dose in patients with neuropathic pain associated with leprosy compared to placebo on the Visual Analogic Scale (VAS) (range 100mm- minimum 0 and maximum 100)

SECONDARY OUTCOMES:
Neuropathic pain | 63 days (9 weeks)
  DN4 (douleur neuropathique 4) + (≥ 4/10)
Neuropathic Pain Symptoms | 63 days (9 weeks)
  To assess the effectiveness of amitriptyline on the reduction of painful symptoms, and on neuropathic dimensions evaluated by the NPSI questionnaire (minimum 0 and maximum 100)
Mensure Quality of Life | 63 days (9 weeks)
  To assess the impact of amitriptyline on the patient's quality of life, depressive and anxiety symptoms, quality of sleep, through the WHOQOL questionnaire (range 0 to 100).
Number of participants with treatment-related adverse events | 63 days (9 weeks)
  To evaluate the number of participants with treatment-related adverse events as assessed by CTCAE v4.03 score 0/1 vs 2/3/4
Predictive factor of response | 63 days (9 weeks)
  assess whether pain phenotype A (NPSI baseline score <15) responded differently to the active drug compared to phenotype B (NPSI score at baseline ≥ 15)
Use of backup pain medication | 63 days (9 weeks)
  To assess the difference in dosage of rescue medication (tramadol) between both treatment arms, by counting the number of pills of tramadol used by each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Andrade, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital Das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No